CLINICAL TRIAL: NCT07005843
Title: A Prospective Multicenter Trial to Evaluate the Elana Anastomotic System for Multi-Arterial Coronary Artery Bypass Grafting
Brief Title: A Study Testing the Elana Device for Multi-Artery Heart Bypass Surgery
Acronym: MULTI-CAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AMT Medical BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MULTI-CAB; NL-009777 (Other: The Central Committee on Research Involving Human Subjects (CCMO))
Record Dates: First submitted 2025-05-26; First posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Bypass Grafting (CABG) Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will receive two or three bypasses using the Elana Anastomotic System. (Experimental): The Elana Anastomotic System is a medical device and is intended to create a suture less blood vessel anastomosis in Coronary Artery Bypass Grafting (CABG) procedures on the beating heart, without blood flow occlusion.
  Interventions: Device: The Elana Anastomotic System

INTERVENTIONS:
Device: The Elana Anastomotic System — The Elana Anastomotic System is a medical device and is intended to create a suture less blood vessel anastomosis in Coronary Artery Bypass Grafting (CABG) procedures on the beating heart, without blo

SUMMARY:
The purpose of the trial is to evaluate the feasibility and safety of multiple Elana Anastomotic Systems to anastomose multiple arterial grafts during coronary artery bypass grafting (CABG). In the first trial performed with the Elana Anastomotic System, the SAFE-CAB trial, only a single anastomosis with the left internal mammary artery (LIMA) was created with the system to the left anterior descending (LAD) coronary artery or a large Diagonal side-branch of the LAD. This is the most important bypass for patients, often described as the anastomosis that guarantees the survival of patients.

However, often multiple anastomoses need to be created during bypass surgery. In the previous study, those anastomoses were performed using vein grafts with standard-of-care hand-sewn techniques. A large body of evidence exists indicating that arterial grafts provide better long-term outcomes for patients undergoing CABG procedures, mainly using the right internal mammary artery (RIMA), but also the Radial Artery, for anastomosis to the Circumflex (Cx) artery and sometimes the Right Coronary Artery. With assurance of safety and effectiveness of the Elena Anastomotic System for LIMA-to-LAD anastomoses and the similarity of the LIMA-to-LAD anastomosis to other arterial anastomoses (e.g., RIMA-to-Cx and RA-to-RCA) as a result of similar vessel diameters and anatomical features, the Elana Anastomotic System is considered to be suitable for multi-arterial bypass procedures.

Therefore, this study aims to expand on the evidence of using the Elana Anastomotic System in a more complete multi-arterial CABG operation, where two or three anastomoses will be created with the Elana Anastomotic System in order to present a more comprehensive solution.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide voluntary written Informed Consent and sign the Informed Consent Form to participate in the study prior to any study-related procedure,
2. Is 18 years or older,
3. Assigned for CABG by the cardiologist and/or cardiothoracic surgeon with one or more vessel disease requiring multiple distal anastomoses, including one on the left anterior descending coronary artery (LAD),
4. Agrees to attend all follow-up assessments for up to 2 years and is willing to comply with specified follow-up evaluations at clinical investigational sites and/or obtain all protocol-specified diagnostic tests.

Exclusion Criteria:

1. Patient is unlikely to cooperate or is legally incompetent, including patients who are institutionalized by court or official order,
2. Any condition which could interfere with the patient's ability to comply with the study,
3. Ongoing participation in any other interventional clinical study,
4. Female patients who are pregnant or lactating,
5. Females who are of child-bearing potential and not taking adequate contraceptive precautions are excluded from the trial. Females of child-bearing potential taking acceptable contraceptive precautions can be included, Note: A highly effective method of birth control and one which is acceptable for this study, is defined as one that can achieve a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence or vasectomized partner.
6. History of cardiothoracic surgery,
7. Active smokers, and smokers who have stopped smoking for less than 1 year,
8. Patients with left ventricular ejection fraction (LVEF)<30%,
9. Concomitant cardiothoracic procedures (i.e. rhythm, aortic, valve surgery, etc.)
10. Requires a planned therapeutic, interventional, or surgical procedure within 1 month (30 days) before or after the scheduled index procedure,
11. Chronic or acute renal failure requiring renal replacement therapy,
12. Cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 3 months (90 days) prior to scheduled index procedure,
13. History of bleeding disorders or coagulopathies,
14. Contraindicated for internal thoracic artery (ITA) harvesting (i.e. obstruction / aortoiliac occlusive disease / radiation therapy at the thoracic region). For additional radial artery harvesting, a negative Allen test is contraindicated,
15. Need for urgent and/or emergent surgery for any reason,
16. During the operation, patients can still be excluded from the study in accordance to the instructions of use for the Elana Anastomotic System.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is defined as the proportion of patients free from all Major Adverse Cardiac Events (MACEs) | Collected 1 year (365 days) after the surgery
  MACE is a composite safety parameter that includes the following events:
  * Cardiac-related mortality,
  * Myocardial Infarction (in the vessel anastomosed with the Elana Anastomotic System)
  * Repeated clinically-driven target-vessel coronary revascularization (in the vessel anastomosed with the Elana Anastomotic System).

SECONDARY OUTCOMES:
The secondary effectiveness endpoint is defined as the graft patency for the ELANA graft/anastomosis. | Performed half an year after the surgery (180 days)
  Graft patency for the ELANA graft/anastomosis will be determined for each ELANA anastomosis separately with coronary angiography (CAG) or coronary computed tomography angiography (CCTA), preferably a photon-counting CT (PCCT).

CONTACTS AND LOCATIONS:
Locations (1):
- St. Antonius Ziekenhuis, Nieuwegein, The Netherlands, Netherlands